CLINICAL TRIAL: NCT06496503
Title: Effect of a School Intervention With Physical Activity on Executive Functions and Relationships With Cardiorespiratory Fitness and Motor Coordination: Randomized Clinical Trial
Brief Title: Effect of a School Intervention With Physical Activity on Executive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Londrina (Other)
Responsible Party: Principal Investigator, Carla Cristiane Silva, Principal Investigator, State University of Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UEL
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy Lifestyle
Keywords: cognitive function; child; physical activity; schoolchildren
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomization will be performed carefully following the recommendations proposed by the Cochrane Collaboration. The process will consist of two stages, firstly, the generation of numbers using a random number table, and secondly, allocation concealment, using opaque, sealed envelopes. After signing the consent form, an envelope will be opened for each child and they will be instructed as to which group they have been allocated, the experimental or control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The team of evaluators, teachers, and researchers who process the results will be completely independent. At all stages of the study (baseline until follow-up) the same outcome assessors will be recruited. None of the individuals, researchers, or evaluators involved will have knowledge as to group allocation. The professional responsible for the physical activities will be hired for this purpose and not belong to the project research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The children included in the experimental group will undergo 12 weeks of physical activity sessions, and it is mandatory that all children complete a minimum of two weekly sessions of physical activity for 50-60 minutes. The activities will consist of content such as motor and cognitive games, sports, dance, and gymnastics. The intensity of the sessions will be checked using accelerometry. The physical activity protocol is adapted from a previously described protocol (CMSP, 2021; Klem, Filha, Monteiro, 2017; Mazzoccante et al.; 2020; Paiano, 2019; Rodrigues, 2018; Rosini et al., 2014). Acceptance of the exercise program in the pediatric population has been previously observed in a pilot study.
  Interventions: Behavioral: Physical activity Protocol
- Control group (No Intervention): The children will follow their usual school routines, including Physical Education classes as part of the curriculum

INTERVENTIONS:
Behavioral: Physical activity Protocol — The children included in the experimental group will undergo 12 weeks of physical activity sessions, and it is mandatory that all children complete a minimum of two weekly sessions of physical activity for 50-60 minutes. The activities will consist of content such as motor and cognitive games, sports, dance, and gymnastics. The intensity of the sessions will be checked using accelerometry. The physical activity protocol is adapted from a previously described protocol (CMSP, 2021; Klem, Filha, Monteiro, 2017; Mazzoccante et al.; 2020; Paiano, 2019; Rodrigues, 2018; Rosini et al., 2014). Acceptance of the exercise program in the pediatric population has been previously observed in a pilot study.
  Arms: Experimental group

SUMMARY:
Previous studies have indicated the relationship between physical activity and cognitive performance, with movement being a promising tool for improving executive functions, especially during childhood, which is a period of intense brain development. Thus, the objective of this project is to verify a school physical activity intervention on executive functions and the relationships with cardiorespiratory fitness and motor coordination. This will be a randomized control trial in accordance with the Consort - Statement, including 118 children of both sexes; 60 in an experimental group and 58 in a control group. The children will follow their usual school routines, including Physical Education classes as part of the curriculum. The experimental group will also participate in an intervention for 12 weeks after school. The intervention will include three weekly physical exercise sessions, lasting between 50 and 60 minutes. The sessions will consist of activities involving games, sports, dance with a focus on aspects of motor coordination and cardiorespiratory fitness, as well as cognitive games. Assessments will be carried out at baseline, after 12 weeks of intervention and after the follow-up period. The students will undergo measurements of body mass and height, as well as nutritional classification using the body mass index (BMI). Following this, a general motor coordination test (KTK), a cardiorespiratory aptitude test (Léger), and tests to assess executive functions (Stroop and Corsi Block) will be applied. Data distribution will be verified using the Shapiro-Wilk's test. The comparisons between different moments (baseline, after 12 weeks, and at follow-up) will be performed using repeated measures ANOVA. Sphericity will be checked by Mauchly's test followed by the Greenhouse- Geisser correction when necessary. To identify differences, the Bonferroni correction will be applied. The significance level will be set at 5% (P<0.05).

DETAILED DESCRIPTION:
During childhood, cognitive aspects of the prefrontal cortex are in the maturation phase. This process is associated with improvements in executive functions, in a continuous process, and although differentiated by its multiple aspects, it seems to correspond with the development peaks of the prefrontal cortex, which occur between 7 and 9 years of age. In addition to the biological alterations arising from the growth and development of the brain, physical activity performed regularly indicates a simple and effective way to improve the executive functions of children. Contreras-Osorio and colleagues stated that physical activity performed at moderate and vigorous intensities is positively related to working memory, reaction time, executive attention, cognitive flexibility, and planning in children and adolescents aged 10 to 12 years. Other authors highlight that activities involving cardiorespiratory fitness and motor coordination provide an increase in cognitive performance, with improvements in planning capacity, memory, self-control, and value judgment, among other fundamental components for social interaction and academic performance In a previous study, Visier-Alfonso and colleagues evaluated 186 school-age children aged 9 to 11 years and demonstrated positive effects on cardiorespiratory fitness, with increased physical activity, and positive changes in inhibitory control, working memory, and brain structure. Additionally, good levels of motor coordination are associated with complex movements and sport-specific skills, and are also essential for the development of higher levels of cognitive function. The relationships between motor skills and executive functions during childhood are based on coactivation events between the prefrontal cortex, the cerebellum, and the basal ganglia during different motor and cognitive tasks, especially when the task is complex, is a new task, or requires speed and concentration. This is because neural regions typically associated with cognitive operations can also be recruited during the performance of motor tasks.

ELIGIBILITY:
Inclusion Criteria:

Healthy

Neurotypical.

Exclusion Criteria:

Clinical or historical of cardiovascular disease

Hypertension

Insulin-dependent diabetes mellitus

Neurodiversity

Not be taking any drugs

Cannot participated in sports practices

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Executive Functions | Will be assessed pre-protocol, after 12 weeks, and 8 weeks after the end of the intervention.
  The executive functions will be assessed pre-protocol, after 12 weeks, and 8 weeks after the end of the intervention (follow-up period). Executive functions will be investigated in the domains of working memory, using the Corsi Block Test (Corsi, 1972; Kessels et al., 2000), and inhibitory control, investigated by the Stroop Test (Stroop, 1935; MacLeod, 1991). For both tests there will be familiarization and reproducibility of measurements for both the children and evaluator. The evaluation will be carried out by a single evaluator blind to group allocation.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Will be assessed pre-protocol, after 12 weeks, and 8 weeks after the end of the intervention.
  The test will be conducted in the field with cones at a distance of 20 meters and a pre-recorded audio track to indicate the speed of each stage. The first stage starts at 8.5 km/h, with an increase of 0.5 km/h every minute, which indicates a change of stage. The test is considered to end when the child is unable to maintain the imposed speed or complete a stage with less than two errors (Léger et al., 1998).
  The prescription of training will be dependent on the individual results for each child based on the last stage completed in the progressive test. At baseline, two field tests will be performed, the first one being a familiarization test and the second being considered as the value prior to the training. In addition, reproducibility of measurements will be tested to indicate the reliability of the results.

OTHER OUTCOMES:
Motor Coordination | Will be assessed pre-protocol, after 12 weeks, and 8 weeks after the end of the intervention.
  To evaluate general motor coordination, the Körperkoordinationstest Für Kinder (KTK) test will be applied (Kiphard; Schiling, 1974, apud Moreira et al., 2019; Nascimento et al., 2019). For all tests involving the KTK battery, there will be familiarization and reproducibility of measurements for both children and the evaluator. The evaluation will be carried out by a single evaluator blind to group allocation.

CONTACTS AND LOCATIONS:
Locations (1):
- School, Nova Fátima, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contreras-Osorio F, Guzman-Guzman IP, Cerda-Vega E, Chirosa-Rios L, Ramirez-Campillo R, Campos-Jara C. Effects of the Type of Sports Practice on the Executive Functions of Schoolchildren. Int J Environ Res Public Health. 2022 Mar 24;19(7):3886. doi: 10.3390/ijerph19073886. PMID 35409571
- [Background] Davis CL, Tomporowski PD, McDowell JE, Austin BP, Miller PH, Yanasak NE, Allison JD, Naglieri JA. Exercise improves executive function and achievement and alters brain activation in overweight children: a randomized, controlled trial. Health Psychol. 2011 Jan;30(1):91-8. doi: 10.1037/a0021766. PMID 21299297
- [Background] de Greeff JW, Bosker RJ, Oosterlaan J, Visscher C, Hartman E. Effects of physical activity on executive functions, attention and academic performance in preadolescent children: a meta-analysis. J Sci Med Sport. 2018 May;21(5):501-507. doi: 10.1016/j.jsams.2017.09.595. Epub 2017 Oct 10. PMID 29054748
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Diamond A, Lee K. Interventions shown to aid executive function development in children 4 to 12 years old. Science. 2011 Aug 19;333(6045):959-64. doi: 10.1126/science.1204529. PMID 21852486
- [Background] Evenson KR, Catellier DJ, Gill K, Ondrak KS, McMurray RG. Calibration of two objective measures of physical activity for children. J Sports Sci. 2008 Dec;26(14):1557-65. doi: 10.1080/02640410802334196. PMID 18949660
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fuster JM. The prefrontal cortex--an update: time is of the essence. Neuron. 2001 May;30(2):319-33. doi: 10.1016/s0896-6273(01)00285-9. No abstract available. PMID 11394996
- [Background] Kessels RP, van Zandvoort MJ, Postma A, Kappelle LJ, de Haan EH. The Corsi Block-Tapping Task: standardization and normative data. Appl Neuropsychol. 2000;7(4):252-8. doi: 10.1207/S15324826AN0704_8. PMID 11296689
- [Background] Leger LA, Mercier D, Gadoury C, Lambert J. The multistage 20 metre shuttle run test for aerobic fitness. J Sports Sci. 1988 Summer;6(2):93-101. doi: 10.1080/02640418808729800. PMID 3184250
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Moreira JPA, Lopes MC, Miranda-Junior MV, Valentini NC, Lage GM, Albuquerque MR. Korperkoordinationstest Fur Kinder (KTK) for Brazilian Children and Adolescents: Factor Analysis, Invariance and Factor Score. Front Psychol. 2019 Nov 19;10:2524. doi: 10.3389/fpsyg.2019.02524. eCollection 2019. PMID 31803092
- [Background] Nascimento WMD, Henrique NR, Marques MDS. KTK MOTOR TEST: REVIEW OF THE MAIN INFLUENCING VARIABLES. Rev Paul Pediatr. 2019 Jun 19;37(3):372-381. doi: 10.1590/1984-0462/;2019;37;3;00013. eCollection 2019. PMID 31241688
- [Background] Serrien DJ, Ivry RB, Swinnen SP. The missing link between action and cognition. Prog Neurobiol. 2007 Jun;82(2):95-107. doi: 10.1016/j.pneurobio.2007.02.003. Epub 2007 Feb 23. PMID 17399884
- [Background] Rigoli D, Piek JP, Kane R, Oosterlaan J. Motor coordination, working memory, and academic achievement in a normative adolescent sample: testing a mediation model. Arch Clin Neuropsychol. 2012 Nov;27(7):766-80. doi: 10.1093/arclin/acs061. Epub 2012 Jul 9. PMID 22777140
- [Background] Roebers CM, Kauer M. Motor and cognitive control in a normative sample of 7-year-olds. Dev Sci. 2009 Jan;12(1):175-81. doi: 10.1111/j.1467-7687.2008.00755.x. PMID 19120425
- [Background] van der Fels IM, Te Wierike SC, Hartman E, Elferink-Gemser MT, Smith J, Visscher C. The relationship between motor skills and cognitive skills in 4-16 year old typically developing children: A systematic review. J Sci Med Sport. 2015 Nov;18(6):697-703. doi: 10.1016/j.jsams.2014.09.007. Epub 2014 Sep 21. PMID 25311901
- [Background] Visier-Alfonso ME, Alvarez-Bueno C, Sanchez-Lopez M, Cavero-Redondo I, Martinez-Hortelano JA, Nieto-Lopez M, Martinez-Vizcaino V. Fitness and executive function as mediators between physical activity and academic achievement. J Sports Sci. 2021 Jul;39(14):1576-1584. doi: 10.1080/02640414.2021.1886665. Epub 2021 Feb 21. PMID 33612080
- [Background] Wassenberg R, Feron FJ, Kessels AG, Hendriksen JG, Kalff AC, Kroes M, Hurks PP, Beeren M, Jolles J, Vles JS. Relation between cognitive and motor performance in 5- to 6-year-old children: results from a large-scale cross-sectional study. Child Dev. 2005 Sep-Oct;76(5):1092-103. doi: 10.1111/j.1467-8624.2005.00899.x. PMID 16150004